CLINICAL TRIAL: NCT04387461
Title: A Phase 2, Single Arm Study of CG0070 Combined With Pembrolizumab in Patients With Non Muscle Invasive Bladder Cancer (NMIBC) Unresponsive to Bacillus Calmette-Guerin (BCG)
Brief Title: Study of CG0070 Given in Combination With Pembrolizumab, in Non-Muscle Invasive Bladder Cancer, Unresponsive to Bacillus Calmette-Guerin
Acronym: CORE-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CG Oncology, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG2003C; KEYNOTE-935 (Other: Merck Sharp & Dohme LLC); MK-3475-935 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: high-grade Ta papillary disease; high-grade T1 papillary disease; carcinoma in situ; Bacillus-Calmette-Guerin Unresponsive
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ | interventions — pembrolizumab; dodecyl maltoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): CG0070 will be administered intravesically (IVE) following a sequence of bladder washes with 5% DDM and normal saline. CG0070 will be administered weekly x 6 on Day 1 to Week 6. If the patient shows persistent high-grade disease at Week 13, the patient will receive another cycle of 6 weekly treatments. If there is no disease present at Week 13 (e.g., complete response) then the patient will receive 3 weekly treatments.
  Beginning at Week 25, patients will receive weekly x 3 treatments every 3 months through Week 49 then every 24 weeks thereafter.
  Pembrolizumab will be given intravenous (IV) concurrently starting on Day 1 and continue every 6 weeks for up to 2 years.
  Interventions: Biological: CG0070; Biological: Pembrolizumab Injection; Other: n-dodecyl-B-D-maltoside

INTERVENTIONS:
Biological: CG0070 — Engineered Oncolytic Adenovirus
Biological: Pembrolizumab Injection — Immune checkpoint inhibitor, Monoclonal antibody
  Other Names: KEYTRUDA®
Other: n-dodecyl-B-D-maltoside — Transduction-enhancing agent.
  Other Names: DDM

SUMMARY:
To evaluate the activity of intravesical administration of CG0070 and intravenous administration of Pembrolizumab in patients with tissue pathology-confirmed non-muscle invasive bladder cancer (NMIBC) who have Bacillus-Calmette-Guerin (BCG) unresponsive disease with carcinoma in situ (CIS) with or without Ta/T1 papillary disease.

DETAILED DESCRIPTION:
An opened label trial designed to evaluate CG0070 and DDM in combination with Pembrolizumab in patients with NMIBC who have failed prior BCG therapy.

The target population of 37 subjects with CIS with or without concomitant high-grade Ta or T1 papillary disease will be enrolled.

BCG failure is defined as persistent or recurrent disease within 12 months of completion of adequate BCG therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Pathologically confirmed NMIBC with CIS (with or without Ta/T1 disease)
* Unresponsive to prior BCG therapy (Lerner 2015) defined as persistent or recurrent CIS alone or with recurrent Ta/T1 (noninvasive papillary disease/tumor invades the sub- epithelial connective tissue) disease within 12 months of completion of adequate BCG therapy. An assessment within 15 months can also qualify when no assessment was performed within 12 months after completion of adequate BCG therapy.

  * Adequate BCG is defined as at least 5 treatments with induction BCG followed by at least 2 BCG treatments as reinduction or maintenance
* Ineligible for radical cystectomy or refusal of radical cystectomy
* Adequate organ function

Key Exclusion Criteria:

* Immuno-deficient due to chronic steroid or other immunosuppressant use, HIV, or prior organ transplant
* Prior treatment with adenovirus-based cancer therapy
* Prior therapy with or intolerant to prior checkpoint inhibitor therapy
* Clinically significant or active cardiac disease
* Active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Complete response rate in patients | 12 months
  Percentage of patients with a complete response as defined by FDA guidance document dated February 2018 for NMIBC.

SECONDARY OUTCOMES:
Incidence of adverse events when CG0070 administered intravesically when combined with pembrolizumab. | 12 months
  Percentage of patients with adverse events by grade as determined by NCI CTCAE v5.0
Median duration of response (DoR) | 12 months
  Median duration of response in patients with a CR or PR
Median overall survival (OS) | 12 months
  Median overall survival in months in patients
Median progression free survival | 12 months
  Median duration of progression free survival of patients

CONTACTS AND LOCATIONS:
Locations (19):
- United States (13):
  - University of California - San Diego, La Jolla, California
  - University of California - Irvine, Orange, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Tampa, Florida
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - Chesapeake Urology, Hanover, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - New York University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Ohio State University, Columbus, Ohio
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Spokane Urology, Spokane, Washington
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Sinchŏn-dong
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li R, Shah PH, Stewart TF, Nam JK, Bivalacqua TJ, Lamm DL, Uchio EM, Geynisman DM, Jacob JM, Meeks JJ, Dickstein R, Pearce SM, Kang SH, Jung SI, Kamat AM, Burke JM, Keegan KA, Steinberg GD. Oncolytic adenoviral therapy plus pembrolizumab in BCG-unresponsive non-muscle-invasive bladder cancer: the phase 2 CORE-001 trial. Nat Med. 2024 Aug;30(8):2216-2223. doi: 10.1038/s41591-024-03025-3. Epub 2024 Jun 6. PMID 38844794